CLINICAL TRIAL: NCT02568332
Title: A Phase I Study to Assess the Safety and Immunogenicity of Prime-boost Immunisations With Vaccine Candidates AdCh3NSmut1 and MVA-NSmut in HIV-1 Seropositive HCV-uninfected Adults on Antiretroviral Therapy (ART)
Brief Title: A Study to Assess the Safety of Hep C Vaccine Candidates in HIV Seropositive Individuals
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: GlaxoSmithKline (Industry); ReiThera Srl (Industry); Cantonal Hospital of St. Gallen (Other); St. James's Hospital, Ireland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PEACHI-02
Record Dates: First submitted 2015-09-22; First posted 2015-10-05 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2017-05

CONDITIONS: Hepatitis C Infection
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Group 1 (Experimental): Interventions: AdCh3NSmut1, MVA-NSmut. Administration schedule: 1 dose AdCh3NSmut1 2.5 x 10^10 vp at week 0 and 1 dose MVA-NSmut 2 x 10^8 pfu at week 8.
  Subjects: 20 HIV seropositive individuals
  Interventions: Biological: AdCh3NSmut1; Biological: MVA-NSmut

INTERVENTIONS:
Biological: AdCh3NSmut1 — Genetic vaccine against Hepatitis C virus infection
Biological: MVA-NSmut — Genetic vaccine against Hepatitis C virus infection

SUMMARY:
This study is aimed at assessing the safety of candidate Hepatitis C (Hep C) vaccines AdCh3NSmut1 and MVA-NSmut when administered to Human Immunodeficiency Virus (HIV) seropositive individuals. This study also aims to assess the cellular immune response generated by these vaccines when administered as mentioned above.

DETAILED DESCRIPTION:
Hepatitis C (Hep C) is a common infection. Worldwide, over 180 million people are infected. Hep C is a blood borne viral infection spread through direct contact with the blood of an infected person. People with Hep C frequently have no symptoms and infection can lead to fibrosis (scarring of the liver), liver failure and cancer. Infection with the Hep C virus (HCV) progresses more rapidly to liver damage in Human Immunodeficiency Virus (HIV)-infected individuals.

Researchers at the University of Oxford have developed a novel candidate vaccine against HCV ('NSmut'). This vaccine has been inserted into the carrier viruses Chimpanzee Adenovirus 3 (AdCh3) and modified vaccinia virus Ankara (MVA), both of which have excellent safety records and have been previously tested in people.

However, the objective of this study is to use exploratory immunological assays to assess whether vaccines for Hep C can induce immune responses in HIV positive individuals that are similar in strength to those in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 seropositive adults must satisfy all the following inclusion criteria to be eligible for the study:

  * Aged 18 to 60 years (inclusive)
  * Resident in or near the trial sites for the duration of the vaccination study for the participant
  * Able and willing (in the Investigator's opinion) to comply with all study requirements
  * HIV Viral Load <50 copies/mL at the last routine HIV follow-up visit within the last 9 months prior to inclusion whilst on treatment with an effective ART regimen
  * Willingness to remain on ART for the study duration
  * CD4 cell count above 350 cells/uL
  * Negative HCV serology and negative HCV RNA polymerase chain reaction (PCR) testing
  * For women of child bearing potential, willingness to practise continuous effective contraception during the study and a negative pregnancy test on the day(s) of vaccination. Effective contraception is defined as a contraceptive method with failure rate of less than 1% per year when used consistently and correctly and, when applicable, in accordance with the product label. In subjects on ART, these are:

    * Injectable progestogen
    * Male partner sterilisation prior to the female subject's entry into the study, and this male is the sole partner for that subject
    * Male condom combined with a vaginal spermicide (foam, gel, film, cream or suppository)
    * Intrauterine device or intrauterine system
    * In addition male partners should use condoms until 3 months after the last vaccination
  * Male trial participants with a female partner of child bearing potential should use condoms until 3 months after the last vaccination. In addition, the female partner should use one of the following contraceptive methods, i.e.

    * Oral or injectable hormonal contraception
    * Sterilisation
    * Intrauterine device or intrauterine system
  * Male trial participants with pregnant partners should use condoms until 3 months after the last vaccination
  * Written informed consent

Exclusion Criteria:

* HIV-1 seropositive adults may not enter the study if any of the following exclusion criteria apply:

  * Participation in another research study involving an investigational product in the 30 days preceding enrolment, or planned use during the study period
  * Prior receipt of a recombinant simian or human adenoviral vaccine
  * Clinical, biochemical (abnormal liver synthetic dysfunction defined by an elevated blood prothrombin time or a low blood albumin level), ultrasonographic, FibroscanTM, or liver biopsy (histology) evidence of cirrhosis or portal hypertension
  * Ongoing or recent (<12 months) AIDS defining illness (US Centers for Disease Control and Prevention (CDC) definition)
  * History of allergic disease or reactions likely to be exacerbated by any component of the vaccine, including egg products or gentamicin.
  * History of clinically significant contact dermatitis
  * Any history of anaphylaxis or serious reaction in relation to vaccination
  * Pregnancy, lactation or willingness/intention to become pregnant during the study
  * Known active malignant disease (except basal cell carcinoma of the skin and cervical carcinoma in situ)
  * Current suspected or known injecting drug abuse (except individuals participating in a heroin substitution program without known or suspected concomitant drug abuse). Participants will be counselled regarding the risk of HCV acquisition during the trial.
  * Seropositive for hepatitis B surface antigen (HBsAg)
  * Positive test for Hepatitis C antibody and/or PCR
  * Moderate neutropenia (Absolute neutrophil count of <1,000 cells/uL)
  * Moderate thrombocytopenia (Platelet count <80,000 cells/uL)
  * Anaemia (Haemoglobin <10g/dL)
  * History of pericarditis and/or myocarditis
  * Heart failure (left ventricular ejection fraction <20%) in the patient history or current medical treatment for heart failure.
  * History of immunologically mediated disease (e.g. inflammatory bowel disease, idiopathic thrombocytopenic purpura, lupus erythematosus, autoimmune hemolytic anemia, scleroderma, rheumatoid arthritis requiring more than intermittent nonsteroidal anti-inflammatory medications for management)
  * History of organ transplantation
  * History of severe psychiatric disease, including psychosis and/or depression, characterised by a suicide attempt, hospitalisation for psychiatric disease, or a period of disability as a result of psychiatric disease.
  * History of a significant coagulopathy (i.e. International Normalised Ratio (INR) > 1.3 and/or Activated Partial Thromboplastin Time (APTT) > 1.5 upper limits of normal) or anticoagulant therapy at time of vaccination
  * Receipt of any oral or systemic antineoplastic or immunomodulatory (e.g. oral systemic corticosteroids) treatment or radiation within 24 weeks before Day 0 or the expectation that such treatment will be needed at any time during the study. Topical or inhaled corticosteroid use is allowed.
  * Any other significant disease, disorder or finding, which, in the opinion of the Investigator, may either put the patient at risk because of participation in the study, or may influence the result of the study, or the patient's ability to participate in the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2015-07-21 (Actual); Primary Completion 2017-01-26 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
Safety of administering HCV prime-boost vaccinations to HIV seropositive individuals, as measured by the proportion of participants who develop a grade 3 or 4 local or systemic reaction | From Day 0 until 6 months after the last vaccination

SECONDARY OUTCOMES:
Cellular immune response generated by HCV prime-boost vaccinations in HIV seropositive individuals, as determined by analysing changes in the magnitude or quality of HCV-specific cellular immune responses | From Day 0 until 6 months after the last vaccination
  Immunogenicity determined by analysing changes from baseline in the magnitude or quality of HCV-specific cellular immune responses. The primary outcome measure for immunogenicity will be the development of T cell responses to HCV epitopes, as determined by Interferon (IFN)-ɣ Enzyme-Linked ImmunoSpot (ELISpot) assay.

CONTACTS AND LOCATIONS:
Overall Officials: Lucy Dorrell, Prof, Study Chair — University of Oxford; Ellie Barnes, Prof, Principal Investigator — University of Oxford; Matthias Hoffmann, Dr, Principal Investigator — Cantonal Hospital of St. Gallen; Colm Bergin, Prof, Principal Investigator — St. James's Hospital, Ireland; Pietro Vernazza, Prof, Principal Investigator — Cantonal Hospital of St. Gallen
Locations (2):
- St James's Hospital, Dublin, Ireland
- Kantonsspital St. Gallen, Sankt Gallen, Switzerland